CLINICAL TRIAL: NCT01532700
Title: An Open-Label Phase 2 Study of Ofatumumab (Arzerra) in Combination With Oral GSK2110183 in the Treatment of Relapsed and Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH-GSK2110183-CLL001
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab; GSK2110183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab with GSK2110183 (Experimental)
  Interventions: Drug: Ofatumumab with GSK2110183

INTERVENTIONS:
Drug: Ofatumumab with GSK2110183 — * GSK2110183 125mg OD continuously
  * Ofatumumab 300mg IV first dose, 2000mg weekly x 7 doses, then 2000mg monthly x 4 doses
  Other Names: Arzerra and GSK2110183

SUMMARY:
This is a phase 2, open-label, single institution trial of combination of intravenous (IV) ofatumumab and oral GSK2110183 in patients with relapsed or refractory Chronic Lymphocytic Leukemia (CLL). Patients must have received at least one prior line of therapy containing fludarabine (single-agent or combination therapy). During the initial 6 months Treatment Phase, ofatumumab will be administered weekly for 8 doses, then once every 4 week cycle for an additional 4 doses (dose and schedule identical to the pivotal phase 2 trial) and GSK2110183 will be given daily PO (Treatment Phase). There will be an initial 10 day lead-in with GSK2110183 alone prior to initiation of ofatumumab to allow for evaluation of changes in cell surface expression due to GSK2110183 and for GSK2110183 pharmacokinetic studies (Lead-in Phase). The official Cycle 1 Day 1 will start on the date of first dose of ofatumumab. Cycle duration = 4 weeks. Patients will be assessed for safety, disease assessment, response, and survival on day 1 of each cycle during the Treatment Phase. A formal review of safety data by the Data Safety Monitoring Board (DSMB) after the first 6 patients have completed cycle 1 of the Treatment Phase will be performed before continuing accrual. All patients achieving SD, PR or CR by the end of the Treatment Phase will proceed to the Maintenance Phase. Patients with PD at any time, including by the end of Treatment Phase, will be taken off study. During the Maintenance Phase, single-agent GSK2110183 will be administered daily for a maximum of 12 months (12 cycles). Maximum duration on any study drug is 18 months (18 cycles). During the Follow-up Phase, patients will be assessed for safety, disease assessment, response, and survival every 3 months through month 36 (year 3), or until subsequent CLL therapy or death, whichever comes first. Key indications for study withdrawal are progressive disease, intolerable toxicity, or completion of therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients must fulfill all of the following criteria to be eligible for admission to the study:

  * A confirmed diagnosis of B-cell CLL by IWCLL 2008 criteria (Appendix 1)
  * Patients must have evidence of disease progression as evidenced by rapid doubling of peripheral lymphocyte count, progressive lymphadenopathy or hepatosplenomegaly, worsening anemia or thrombocytopenia, or progressive constitutional symptoms [including fatigue, weight loss, night sweats, fever (without infection)]
  * Must be relapsed or refractory to at least one prior fludarabine-containing regimen (no maximum number of prior regimens).
  * Age > 18 years.
  * ECOG performance status of 0, 1 or 2 (Appendix 3)
  * Signed the Informed Consent form
  * Life expectancy of ≥ 6 months
  * Able to swallow and retain oral medication
  * Normal HbA1C ≤ 0.07
  * Fasting blood sugar < 7mmol/L

Exclusion Criteria:

* Subjects meeting any of the following criteria are excluded from this study:

  * CLL therapy, including stem cell transplantation, within 4 weeks of study initiation. Corticosteroids alone may be administered up to seven days prior to the first dose of study drug.
  * Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study
  * Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to start of therapy
  * Known hypersensitivity to ofatumumab, GSK2110183, or any components therein.
  * Anticoagulants are permitted only if the subject meets PTT and INR entry criteria (INR and PTT ≤ 1.5 times upper normal limit). Their use must be monitored in accordance with local institutional practice.
  * Current use of any anti-platelet agent (e.g. dipyridamole, clopidogrel) other than aspirin (81mg daily).
  * Current use of a prohibited medication based on potential drug-drug interaction - a complete list is found in Appendix 1
  * Known CNS involvement with CLL
  * Transformation to aggressive B-cell malignancy (e.g. large B-cell lymphoma, Richter's syndrome, prolymphocytic leukemia [PLL])
  * "Active" autoimmune disease - prior history of autoimmune hemolysis (DAT positive or negative) or immune thrombocytopenia without current active autoimmune disease is allowed
  * Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable non-hepatitis B or C chronic liver disease per investigator assessment - please see below for Hepatitis B and C criteria)
  * Previously diagnosed diabetes mellitus (Type 1 or 2)
  * Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
  * Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, and tuberculosis.
  * Any medical condition that would require long-term use (> 1 month) of systemic corticosteroids during study treatment (excludes topical or inhaled corticosteroid use)
  * History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
  * QTc ≥ 470 msec on screening ECG
  * Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to study entry, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
  * Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
  * Any major surgery within the prior 4 weeks.
  * Known HIV positive
  * Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
  * Positive serology for hepatitis C (HC) defined as a positive test for HCAb, in which case reflexively perform a HC RIBA immunoblot assay on the same sample to confirm the result
  * Screening laboratory values: platelets ≤ 30 x 109/L,neutrophils ≤ 0.7 x 109/L,creatinine ≥ 2.0 times upper normal limit, total bilirubin ≥ 1.5 times upper normal limit (unless due to a known history of Gilbert's disease), ALT ≥ 2.5 times upper normal limit, alkaline phosphatase ≥ 2.5 times upper normal limit, INR and PTT ≤ 1.5 times upper normal limit
  * Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening.
  * Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as intrauterine device, double barrier method or total abstinence. Oral contraceptives are not adequate due to potential drug-drug interaction.
  * Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chen, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment was stopped as of 13 Sep 2016. 28 patients were enrolled. Data analysis is complete and manuscript has been being submitted.
Groups:
- Ofatumumab With GSK2110183: Ofatumumab with GSK2110183: - GSK2110183 125mg OD continuously
  - Ofatumumab 300mg IV first dose, 2000mg weekly x 7 doses, then 2000mg monthly x 4 doses
Period: Overall Study
Arm/Group | Ofatumumab With GSK2110183
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab With GSK2110183
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate, as Per the IWCLL 2008 Response Criteria
Description: IWCLL Response Criteria 2008-Hallek. Complete response (CR): requires peripheral blood lymphocytes < 4 x 109/L, absence of significant lymphadenopathy (>1.5cm), no organomegaly, normal CBC, bone marrow must be at least normocellular; Complete Remission with incomplete bone marrow recovery (CRi): fulfill all the criteria for CR but have persistent anemia, thrombocytopenia or neutropenia apparently unrelated to disease activity but related to drug toxicity; Partial Remission (PR): ≥ 50% decrease in the peripheral blood lymphocytes from baseline, > 50% reduction in the sum products of up to 6 lymph nodes, > 50% reduction in hepatomegaly and/or neutrophils > 1.5 x109/L, platelets > 100 x109/L, hemoglobin > 110 g/L; Stable Disease: Not CR, PR or PD (equivalent to nonresponse); Progressive Disease: Lymphadenopathy, or appearance of any new lesion/organomegaly, > 50% increase in the size of the liver and/or spleen, > 50% increase in the absolute number of circulating lymphocytes
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab With GSK2110183
Number analyzed (Participants) | 28
Participants
  Complete response | 1
  Partial response | 13
  Stable disease | 14

2. Secondary Outcome: Stable Disease, Response Rate, Toxicity (as Graded Per NCI CTC Version 4.03)
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab With GSK2110183
Number analyzed (Participants) | 28
percentage of participants
  Response rate (%) | 50
  Stable Disease (%) | 50
  Upper respiratory Infections (%) | 71
  Cough (%) | 64
  Diarrhea (%) | 61
  Dyspnea (%) | 36
  Lung Infections (%) | 18
  Upper respiratory infections (%) | 71
  Skin (%) | 32
  Urinary tract infection (%) | 18
  Neutropenia Grade 3-4(%) | 39
  Thrombocytopenia Grade 3-4 (%) | 32
  Anemia Grade 3-4 (%) | 25
  Infusion related reactions (%) | 75

3. Secondary Outcome: Median Progression Free Survival, Overall Survival
Description: Progression Free Survival (PFS) is defined as the length of time between the date of first dose of study treatment (GSK2110183) and the earliest date of disease progression or death due to any cause.
  Overall survival is defined as the length of time between the date of first dose of study treatment (GSK2110183) and death due to any cause.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab With GSK2110183
Number analyzed (Participants) | 28
months
  Median PFS time (months) | 8.5 [7.7 to 13.2]
  1 year overall survival time (months) | 88.3 [76.6 to 100]
  2 year overall survival time | 68.1 [46.0 to 100]

4. Secondary Outcome: Median Duration of Response
Description: Duration of Response (DOR) is defined, for the subset of patients with a CR or PR, as the time from first documented evidence of CR or PR until first documented disease progression or death due to any cause. Duration of response will be summarized descriptively using Kaplan-Meier medians and quartiles.
Time Frame: 36 months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Ofatumumab With GSK2110183
Number analyzed (Participants) | 28
months | 6.4 [3.2 to 11.7]

ADVERSE EVENTS:
Time Frame: Twenty-eight patients were evaluable for toxicity and response from the time of their first dose of afuresertib. Adverse events were graded using NCI Common Toxicity Criteria v4.03 at each visit. Patients were assessed four weeks after study discontinuation. Thereafter, for patients off-study for progressive disease, follow-up documented ongoing/late toxicities and death. For patients off-study with CR, PR, or SD, follow-up was every three months until progression or death.
Arm/Group | Ofatumumab With GSK2110183
All-Cause Mortality (participants affected / at risk) | 27/27
Serious Adverse Events (participants affected / at risk) | 14/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab With GSK2110183 (N=27)
febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Bronchial infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 4
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 2
Back pain ?Progressive CLL (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma of pulmonary origin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive squamous cell carcinoma-malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bilateral hydronephrosis (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Reproductive system and breast disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab With GSK2110183 (N=27)
Infusion related reaction (General disorders) | 20
Fever (General disorders) | 13
Paresthesias (Nervous system disorders) | 7
Fatigue (General disorders) | 8
Dizziness (Nervous system disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 5
leg edema (General disorders) | 4
Dysgeusia (Nervous system disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Dyspepsia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 4
Anemia (Blood and lymphatic system disorders) | 12
Neutropenia (Investigations) | 10
Thrombocytopenia (Investigations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT01532700/Prot_SAP_000.pdf